CLINICAL TRIAL: NCT07371624
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Allogeneic Adipose-Derived Mesenchymal Stromal Cell Injection (B2065) in Participants With Acute Ischemic Stroke.
Brief Title: A Study of the Safety, Tolerability and Preliminary Efficacy of B2065 in Patients With Acute Ischemic Stroke.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSL-BM-B2065-I/IIa
Record Dates: First submitted 2026-01-08; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B2065 (Experimental): Phase I dose escalation includes 5.0×10^7 cells (1 bag), 1.5×10^8 cells (3 bags), and 4.5×10^8 cells (9 bags), formulated in 1% human serum albumin and sodium chloride injection.
  Phase IIa dose expansion will select 1-2 dose cohorts from Phase I. Participants will be randomized in a 2:1 ratio (B2065:placebo).
  Interventions: Drug: B2065
- Placebo (Placebo Comparator): Placebo (1% human serum albumin in sodium chloride injection) administered by intravenous infusion, with matched volume and number of bags.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: B2065 — Administered by intravenous infusion.
  Arms: B2065
Drug: Placebo — Administered by intravenous infusion.
  Arms: Placebo

SUMMARY:
This Phase I/IIa, randomized, double-blind, placebo-controlled study evaluates the safety, tolerability, and preliminary efficacy of B2065, an allogeneic adipose-derived mesenchymal stromal cell (AD-MSC) injection, in patients with acute ischemic stroke. Participants receive a single intravenous infusion of B2065 or placebo within 36 hours of stroke symptom onset. Phase I uses dose escalation with sentinel dosing to assess dose-limiting toxicities within 28 days and to inform dose selection. Phase IIa expands 1-2 selected dose level(s) and randomizes participants 2:1 (B2065:placebo). Safety and functional outcomes are assessed through 24 months.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18 to 75 years (inclusive of the boundary values), with no restriction on sex.
2. Patients with ischemic stroke confirmed by imaging examinations (CT/MRI).
3. Time from onset of stroke symptoms to administration of the investigational product ≤36 hours; for wake-up stroke, the time of onset is defined as the last-known-well time (the last time the patient was observed to be normal).
4. NIHSS score at screening is 8 to 20.
5. The patient or legally authorized representative is willing to participate in this trial and agrees to sign the informed consent form.

Exclusion Criteria

1. Patients who have received intravenous thrombolysis and/or mechanical thrombectomy prior to dosing.
2. Modified Rankin Scale (mRS) score ≥2 before stroke onset.
3. Patients who currently have intracranial hemorrhagic diseases (e.g., intracerebral hemorrhage, epidural hematoma, subarachnoid hemorrhage, etc.), or who have brain tumors, cerebrovascular malformations, multiple sclerosis, a history of severe traumatic brain injury, encephalitis, or other conditions causing stroke-like symptoms.
4. Patients who are unable to undergo CT and/or MRI examinations.
5. Patients with decreased level of consciousness (NIHSS item 1a score ≥2).
6. Patients who may have major neurologic or psychiatric disorders that seriously interfere with the participant's compliance with trial assessments.
7. Body temperature >38°C prior to dosing, and the investigator assesses that there is a risk of infection.
8. Patients with uncontrollable active infection; or patients who have received systemic anti-infective therapy within 7 days prior to dosing and, in the investigator's judgment, may be likely to convert to uncontrollable active infection in the short term.
9. Patients with current or prior severe diseases of other organ systems, including but not limited to:

   1. Patients with severe heart failure (NYHA Class III or IV) and/or severe respiratory failure;
   2. Patients with renal disease with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m²;
   3. Advanced liver disease, such as hepatitis or liver cirrhosis;
   4. Patients positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg); patients positive for hepatitis B e antibody (HBeAb) and/or hepatitis B core antibody (HBcAb) with quantitative HBV-DNA above the upper limit of normal; patients with any of the following test results positive: hepatitis C virus antibody (HCV-Ab), Treponema pallidum antibody (TP-Ab), or human immunodeficiency virus antibody (HIV-Ab);
   5. Patients with hypertension not controlled after taking therapeutic medications, with systolic blood pressure ≥185 mmHg and/or diastolic blood pressure ≥110 mmHg;
   6. Blood glucose <2.8 mmol/L (50 mg/dL) or >22.2 mmol/L (400 mg/dL).
10. Screening laboratory tests meeting any of the following criteria:

    1. Serum alanine aminotransferase (ALT) ≥3× upper limit of normal (ULN);
    2. Serum aspartate aminotransferase (AST) ≥3× ULN;
    3. Serum creatinine (Cr) ≥2× ULN;
    4. Absolute neutrophil count (ANC) <1.5×10^9/L;
    5. Platelet count (PLT) <100×10^9/L;
    6. Hemoglobin (Hgb) <90 g/L;
    7. International normalized ratio (INR) >1.7 or activated partial thromboplastin time (APTT) >1.25× ULN.
11. Patients with malignant tumors or other diseases with an expected survival of less than 2 years.
12. Patients with other acquired or congenital immunodeficiency diseases, or those currently using immunosuppressants.
13. Patients who, upon screening inquiry, have alcohol dependence or a history of drug abuse.
14. Pregnant or breastfeeding women; or those who plan to conceive, donate sperm, or donate oocytes during the trial and/or are unwilling to take effective contraception measures.
15. Patients who participated in any other clinical trial within 1 month prior to screening.
16. Patients who are allergic to any component of the investigational product.
17. Patients deemed by the investigator to be unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with dose-limiting toxicity | Within 28 days after dosing.
  Tolerability assessment (Phase l dose-escalation stage only). Dose-limiting toxicity (DLT) was defined as Grade ≥3 adverse events related to B2065 occurring within 28 days after dosing, assessed according to CTCAE (v6.0).
Infusion reactions | Within 7 days, 14 days, and 28 days.
  Infusion-related reactions include hypersensitivity reactions and systemic complications.
All-cause mortality | Within 14 days,12 months, and 24 months.
Tumorigenicity surveillance | Month 6 and month 24.
  Tumorigenicity assessments included chest and abdominal CT scans and tumor markers, including alpha-fetoprotein (AFP), carcinoembryonic antigen (CEA), carbohydrate antigen 125 (CA125), carbohydrate antigen 19-9 (CA199), squamous cell carcinoma antigen (SCCA), prostate-specific antigen (PSA), and neuron-specific enolase (NSE). Additional tumor markers assessed in female participants included carbohydrate antigen 15-3 (CA15-3), human chorionic gonadotropin (hCG), serum ferritin (SF), and beta-2 microglobulin (β2-MG).
Adverse events (AEs) | Day1 to month 24.
  Occurrence rate of AEs.

SECONDARY OUTCOMES:
Proportion of participants with an modified Rankin Scale score of 0-2 after treatment | Day 28, day 90, month 6, and month 12.
  The modified Rankin Scale (mRS) is used to assess functional recovery after stroke. The scale consists of 7 levels, ranging from 0 (no symptoms) to 6 (death). An mRS score of 0-1 is defined as a favorable clinical outcome, and an mRS score of 0-2 is defined as functional independence. The mRS will be assessed by investigators at screening/baseline, Day 28, Day 90, Month 6, and Month 12.
Proportion of participants with an modified Rankin Scale score of 0-1 after treatment | Day 28, day 90, month 6, and month 12.
  The modified Rankin Scale (mRS) is used to assess functional recovery after stroke. The scale consists of 7 levels, ranging from 0 (no symptoms) to 6 (death). An mRS score of 0-1 is defined as a favorable clinical outcome, and an mRS score of 0-2 is defined as functional independence. The mRS will be assessed by investigators at screening/baseline, Day 28, Day 90, Month 6, and Month 12.
Proportion of participants with a decrease in NIH Stroke Scale score of ≥4 points from baseline or an NIHSS score ≤1 after treatment | 24 hours, day 3, day 7, day 14, and month 12.
  The NIH Stroke Scale (NIHSS) quantitatively evaluates the severity of neurological deficits in stroke patients, with scores ranging from 0 (no deficit) to 42 (most severe deficit). A decrease in NIHSS score of ≥4 points from baseline (or an NIHSS score ≤1) is defined as neurological improvement. The NIHSS will be assessed by investigators at each visit. The NIHSS score assessed within 20 minutes prior to dosing will be used as the baseline value.
Change from baseline in NIH Stroke Scale score after treatment | 24 hours, day 3, day 7, day 14, and month 12.
  The NIH Stroke Scale (NIHSS) quantitatively evaluates the severity of neurological deficits in stroke patients, with scores ranging from 0 (no deficit) to 42 (most severe deficit). A decrease in NIHSS score of ≥4 points from baseline (or an NIHSS score ≤1) is defined as neurological improvement. The NIHSS will be assessed by investigators at each visit. The NIHSS score assessed within 20 minutes prior to dosing will be used as the baseline value.
Proportion of participants with a Barthel Index score of 95-100 after treatment | Day 28, day 90, month 6, and month 12.
  The Barthel Index (BI) is used to evaluate a participant's ability to perform activities of daily living (ADL). It includes 10 items: feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, transfers (bed to chair and back), mobility, and stair climbing. Total scores range from 0 (complete dependence) to 100 (independence). A BI score of 95-100 is defined as slight or no disability.
EQ-5D-5L score after treatment | Day 28, day 90, month 6, and month 12.
  The EQ-5D is a standardized instrument for measuring health status developed by the EuroQol Group, providing a simple and generic measure of health. The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system covers five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems/unable to perform. The EQ VAS is a vertical visual analogue scale anchored by "the best health you can imagine" and "the worst health you can imagine." Participants will select the option that best describes their health state in each dimension and record their self-rated health on the EQ VAS.

OTHER OUTCOMES:
Immune Biomarkers [Exploratory Outcome 1] | Pre-dose (within 20 minutes prior to dosing) and Day 3, Day 28, and Day 90 post-dose.
  Immune Biomarkers (IgG, IgM, IgA, IgE; Treg; TNF-α).
Nerve Growth Factor [Exploratory Outcome 2] | Pre-dose (within 20 minutes prior to dosing) and Day 7, Day 28, Day 90, and Month 12 post-dose.
  Nerve Growth Factor (NGF).
Anti-drug Antibodies [Exploratory Outcome 3] | Pre-dose (within 20 minutes prior to dosing) and Day 14, Day 28, Day 90, and Month 12 post-dose.
  Anti-drug Antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China